CLINICAL TRIAL: NCT02823652
Title: COMET - Communication and Education in Tumor Profiling: A Randomized Study of Pre-Disclosure Genetic Education v. Usual Care in Tumor Profiling for Advanced Cancer and a Pilot Study of Remote Genetic Counseling for Participants With Potential Germline Mutations Identified on Tumor Profiling
Brief Title: Pre-Test Genetic Education and Remote Genetic Counseling in Communicating Tumor Profiling Results to Patients With Advanced Cancer
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: ECOG-ACRIN Cancer Research Group (Network)
Collaborators: National Cancer Institute (NCI) (NIH)
Responsible Party: Sponsor
Organization: Eastern Cooperative Oncology Group (Network)
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Health Services Research
Other Study IDs: EAQ152; NCI-2015-02253 (Registry Identifier: CTRP (Clinical Trial Reporting Program)); EAQ152 (Other: ECOG-ACRIN Cancer Research Group); EAQ152 (Other: CTEP)
Record Dates: First submitted 2016-06-21; First posted 2016-07-06 (Estimated); Results first posted 2024-02-28 (Actual); Last update posted 2024-02-28 (Actual); Status verified 2023-12

CONDITIONS: Advanced Malignant Neoplasm; Locally Advanced Malignant Neoplasm
MeSH Terms: interventions — Counseling; Genetic Counseling; Genetic Testing

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Arm A (Step 1: internet-based intervention) (Experimental): Patients receive web-based genetic education consisting of general information about testing tumors for genetic mutations.
  Interventions: Other: Internet-Based Intervention; Other: Survey Administration
- Arm B (Step 1: usual care control) (Active Comparator): Patients receive standard genetic education consisting of conversations with the treating physicians, interaction with and information from the clinical staff, and information from usual resources about testing for genetic mutations.
  Interventions: Other: standard genetic education; Other: Survey Administration
- Step 2 - genetic counseling (Experimental): Patients who meet the criteria for the remote counseling substudy will receive genetic counseling over the telephone and undergo germline testing.
  Interventions: Other: Genetic Counseling; Other: Genetic Testing; Other: Survey Administration

INTERVENTIONS:
Other: standard genetic education — Undergo usual care
  Other Names: counseling; Counseling Intervention
  Arms: Arm B (Step 1: usual care control)
Other: Genetic Counseling — Complete remote counseling
  Arms: Step 2 - genetic counseling
Other: Genetic Testing — Undergo germline testing
  Other Names: genetic analysis; Genetic Examination; Genetic Test
  Arms: Step 2 - genetic counseling
Other: Internet-Based Intervention — Complete on-line genetic education
  Arms: Arm A (Step 1: internet-based intervention)
Other: Survey Administration — Ancillary studies

SUMMARY:
This research trial studies how well pre-test genetic education and remote genetic counseling works in communicating tumor profiling results to patients with advanced cancer. Web-based genetic education before receiving tumor profiling results and remote genetic counseling for patients with potential germline mutations may increase genetic knowledge and reduce distress for patients with advanced cancer.

DETAILED DESCRIPTION:
PRIMARY OBJECTIVES:

I. To evaluate the efficacy of web-based pre-disclosure genetic education (i.e. before receipt of tumor profile results) to increase knowledge (genetic knowledge and knowledge of test benefits and limitations). (Step 1)

II. To evaluate the efficacy of web-based pre-disclosure genetic education (i.e. before receipt of tumor profile results) to decrease distress (anxiety, depression and cancer specific worry) compared to usual care services in patients undergoing tumor profiling for advanced cancer. (Step 1)

III. To evaluate the uptake of remote genetic counseling (Step 2)

IV. To evaluate the uptake of germline testing among advanced cancer patients with a potential clinically significant incidental germline mutation identified through tumor profiling in the Molecular Analysis for Therapy Choice (MATCH) trial. (Step 2)

SECONDARY OBJECTIVES:

I. To evaluate potential moderators suggested by the self-regulation theory of health behavior (SRTHB) (e.g. test result, sociodemographic factors, health literacy, baseline knowledge or distress) to changes in knowledge of genetic disease and test benefits and limitations. (Step 1)

II. To evaluate potential moderators suggested by the SRTHB (e.g test result, sociodemographic factors, health literacy, baseline knowledge or distress) to changes in distress in patients undergoing tumor profiling for advanced cancer. (Step 1)

III. To evaluate factors associated with uptake of genetic counseling and germline testing. (Step 2)

IV. To evaluate cognitive, affective and behavioral (communication to relatives) responses to confirmatory germline testing in advanced cancer patients with potential clinically significant incidental germline mutation identified in tumor profiling. (Step 2)

OUTLINE:

STEP I (PRIMARY INTERVENTION STUDY): Participants are randomized to 1 of 2 arms.

ARM A: Patients receive web-based genetic education consisting of general information about testing tumors for genetic mutations.

ARM B: Patients receive standard genetic education consisting of conversations with the treating physicians, interaction with and information from the clinical staff, and information from usual resources about testing for genetic mutations.

STEP II (SECONDARY GENETIC COUNSELING SUBSTUDY):

Patients who meet the criteria for the remote counseling substudy will receive genetic counseling over the telephone and undergo germline testing.

After completion of study treatment, patients are followed up periodically.

ELIGIBILITY:
Inclusion Criteria:

* (STEP 1) - PRIMARY INTERVENTION STUDY (RANDOMIZED CONTROLLED TRIAL [RCT]):
* Patients must be registered to the first screening step (Step 0) for the National Cancer Institute (NCI)-MATCH trial (EAY131)
* Patients must speak English and have an adequate ability to view a website (primary intervention study)
* (STEP 2) - SECONDARY GENETIC COUNSELING SUBSTUDY:
* Patients must have a potential germline mutation, as determined by the NCI-MATCH tumor profiling assay
* Patients must be able to speak English and hear by phone

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 601 (Actual)
Dates: Start 2016-10-25 (Actual); Primary Completion 2019-12-26 (Actual); Study Completion 2019-12-26 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Angela Bradbury, Principal Investigator — ECOG-ACRIN Cancer Research Group
Locations (1):
- ECOG-ACRIN Cancer Research Group, Philadelphia, Pennsylvania, United States

REFERENCES:
- [Derived] Bradbury AR, Lee JW, Gaieski JB, Li S, Gareen IF, Flaherty KT, Herman BA, Domchek SM, DeMichele AM, Maxwell KN, Onitilo AA, Virani S, Park S, Faller BA, Grant SC, Ramaekers RC, Behrens RJ, Nambudiri GS, Carlos RC, Wagner LI. A randomized study of genetic education versus usual care in tumor profiling for advanced cancer in the ECOG-ACRIN Cancer Research Group (EAQ152). Cancer. 2022 Apr 1;128(7):1381-1391. doi: 10.1002/cncr.34063. Epub 2021 Dec 10. PMID 34890045

RESULTS

PARTICIPANT FLOW:
Recruitment Details: A total of 601 patients were enrolled between October 25, 2016 and March 31, 2019.
Groups:
- Arm A (Step 1: Internet-based Intervention; Step 2: Genetic Counseling Substudy): Patients receive web-based genetic education consisting of general information about testing tumors for genetic mutations.
  Patients who meet the criteria for the remote counseling substudy will receive genetic counseling over the telephone and undergo germline testing in Step 2. Not all patients in Step 1 will be eligible and willing to participate in Step 2.
- Arm B (Step 1: Usual Care Control; Step 2: Genetic Counseling Substudy): Patients receive standard genetic education consisting of conversations with the treating physicians, interaction with and information from the clinical staff, and information from usual resources about testing for genetic mutations.
  Patients who meet the criteria for the remote counseling substudy will receive genetic counseling over the telephone and undergo germline testing in Step 2. Not all patients in Step 1 will be eligible and willing to participate in Step 2.
- Arm C (Step 1: no Participation; Step 2: Genetic Counseling Substudy): These are patients who did not participate in the primary on-line genetic education study (Step 1) but meet the criteria for the remote counseling substudy. These patients will receive genetic counseling over the telephone and undergo germline testing in Step 2.
Period: Step 1: On-line Genetic Education Study
Arm/Group | Arm A (Step 1: Internet-based Intervention; Step 2: Genetic Counseling Substudy) | Arm B (Step 1: Usual Care Control; Step 2: Genetic Counseling Substudy) | Arm C (Step 1: no Participation; Step 2: Genetic Counseling Substudy)
Started | 293 | 301 | 7
Baseline Survey Completion | 235 | 237 | 0
Completed | 235 | 237 | 0
Not Completed | 58 | 64 | 7
Not completed — Baseline survey not done | 58 | 64 | 7
Period: Step 2: Genetic Counseling Substudy
Arm/Group | Arm A (Step 1: Internet-based Intervention; Step 2: Genetic Counseling Substudy) | Arm B (Step 1: Usual Care Control; Step 2: Genetic Counseling Substudy) | Arm C (Step 1: no Participation; Step 2: Genetic Counseling Substudy)
Started | 9 | 4 | 7
Eligible Patients | 7 | 4 | 7
Completed | 3 | 2 | 5
Not Completed | 6 | 2 | 2
Not completed — Ineligible | 2 | 0 | 0
Not completed — Withdrawal by Subject | 2 | 0 | 1
Not completed — Other | 2 | 2 | 1

BASELINE CHARACTERISTICS:
Population: All patients enrolled on this study
Groups:
- Arm A (Step 1: Internet-based Intervention; Step 2: Genetic Counseling Substudy): Patients receive web-based genetic education consisting of general information about testing tumors for genetic mutations.
  Patients who meet the criteria for the remote counseling substudy will receive genetic counseling over the telephone and undergo germline testing in Step 2.
- Arm B (Step 1: Usual Care Control; Step 2: Genetic Counseling Substudy): Patients receive standard genetic education consisting of conversations with the treating physicians, interaction with and information from the clinical staff, and information from usual resources about testing for genetic mutations.
  Patients who meet the criteria for the remote counseling substudy will receive genetic counseling over the telephone and undergo germline testing in Step 2.
- Arm C (Step 1: no Participation; Step 2: Genetic Counseling Substudy): Patients who did not participate in the primary on-line genetic education study (Step 1) but meet the criteria for the remote counseling substudy. These patients will receive genetic counseling over the telephone and undergo germline testing in Step 2.
- Total: Total of all reporting groups
Arm/Group | Arm A (Step 1: Internet-based Intervention; Step 2: Genetic Counseling Substudy) | Arm B (Step 1: Usual Care Control; Step 2: Genetic Counseling Substudy) | Arm C (Step 1: no Participation; Step 2: Genetic Counseling Substudy) | Total
Number analyzed (Participants) | 293 | 301 | 7 | 601
Age, Continuous [Median (Full Range); unit: years] | 65 [27 to 85] | 65 [33 to 91] | 62 [42 to 77] | 65 [27 to 91]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 161 | 168 | 6 | 335
  Male | 132 | 133 | 1 | 266
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 2 | 6 | 0 | 8
  Not Hispanic or Latino | 286 | 291 | 6 | 583
  Unknown or Not Reported | 5 | 4 | 1 | 10
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 1 | 0 | 0 | 1
  Asian | 4 | 3 | 0 | 7
  Native Hawaiian or Other Pacific Islander | 1 | 1 | 0 | 2
  Black or African American | 12 | 16 | 1 | 29
  White | 268 | 274 | 6 | 548
  More than one race | 1 | 1 | 0 | 2
  Unknown or Not Reported | 6 | 6 | 0 | 12

OUTCOME MEASURES:

1. Primary Outcome: Change of Scores on Cancer Genetic Knowledge Scale From Baseline to Post-genetic Education
Description: There are 14 items in the questionnaire of Cancer Genetic Knowledge Scale. The total score ranges between 14 and 70. Higher scores indicate more/better knowledge. The questionnaire was administered at baseline and post-genetic education. The change of scores from baseline to post-genetic education were calculated and compared between the two arms (arms A and B) at Step 1.
Time Frame: Assessed at baseline and post-genetic education (about 1-2 weeks post-baseline)
Population: Eligible patients who completed both baseline and post-genetic education questionnaires were included in the analysis.
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Arm A (Step 1: Internet-based Intervention) | Arm B (Step 1: Usual Care Control)
Number analyzed (Participants) | 184 | 178
score on a scale | 1.43 (4.31) | -0.80 (3.63)
Statistical Analysis 1: Comparison: Arm A (Step 1: Internet-based Intervention) vs Arm B (Step 1: Usual Care Control); Test type: Superiority; p < .0001, t-test, 2 sided

2. Primary Outcome: Change of Scores on Patient-Reported Outcomes Measurement Information System (PROMIS) - Depression From Baseline to Post-genetic Education
Description: There are 4 items in the PROMIS - Depression questionnaire. The total score ranges between 4 and 20. Higher scores indicate more depression. The questionnaire was administered at baseline and post-genetic education. The change of scores from baseline to post-genetic education were calculated and compared between the two arms (arms A and B) at Step 1.
Time Frame: Assessed at baseline and post-genetic education (about 1-2 weeks post-baseline)
Population: Eligible patients who completed both baseline and post-genetic education questionnaires were included in the analysis.
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Arm A (Step 1: Internet-based Intervention) | Arm B (Step 1: Usual Care Control)
Number analyzed (Participants) | 195 | 193
score on a scale | 0.23 (2.36) | -0.30 (2.48)
Statistical Analysis 1: Comparison: Arm A (Step 1: Internet-based Intervention) vs Arm B (Step 1: Usual Care Control); Test type: Superiority; p = 0.035, t-test, 2 sided

3. Primary Outcome: Change of Scores on Patient-Reported Outcomes Measurement Information System (PROMIS) - Anxiety From Baseline to Post-genetic Education
Description: There are 4 items in the PROMIS - Anxiety questionnaire. The total score ranges between 4 and 20. Higher scores indicate more anxiety. The questionnaire was administered at baseline and post-genetic education. The change of scores from baseline to post-genetic education were calculated and compared between the two arms (arms A and B) at Step 1.
Time Frame: Assessed at baseline and post-genetic education (about 1-2 weeks post-baseline)
Population: Eligible patients who completed both baseline and post-genetic education questionnaires were included in the analysis.
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Arm A (Step 1: Internet-based Intervention) | Arm B (Step 1: Usual Care Control)
Number analyzed (Participants) | 202 | 201
score on a scale | -0.32 (2.33) | -0.55 (2.24)
Statistical Analysis 1: Comparison: Arm A (Step 1: Internet-based Intervention) vs Arm B (Step 1: Usual Care Control); Test type: Superiority; p = 0.312, t-test, 2 sided

4. Primary Outcome: Change of Scores on Impact of Events Scale (IES) From Baseline to Post-genetic Education
Description: There are 14 items in the questionnaire of Impact of Events Scale (IES). The total score ranges between 0 and 70. Higher scores indicate more stress. The questionnaire was administered at baseline and post-genetic education. The change of scores from baseline to post-genetic education were calculated and compared between the two arms (arms A and B) at Step 1.
Time Frame: Assessed at baseline and up to 14 days post-baseline
Population: Eligible patients who completed both baseline and post-genetic education questionnaires were included in the analysis.
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Arm A (Step 1: Internet-based Intervention) | Arm B (Step 1: Usual Care Control)
Number analyzed (Participants) | 183 | 191
score on a scale | -1.79 (9.43) | -0.19 (9.86)
Statistical Analysis 1: Comparison: Arm A (Step 1: Internet-based Intervention) vs Arm B (Step 1: Usual Care Control); Test type: Superiority; p = 0.11, t-test, 2 sided

5. Primary Outcome: Proportion of Participants Who Complete Remote Genetic Counseling in the Genetic Counseling Substudy (Step 2)
Description: Among participants who registered in the genetic counseling substudy (Step 2), the proportion of participants who completed remote genetic counseling will be reported. The proportion is defined as "the number of participants who completed remote genetic counseling divided by the number of participants who agreed to participate in the genetic counseling study".
Time Frame: Assessed at baseline at Step 2
Population: Eligible patients who agreed to participate in Step 2 genetic counseling substudy
Measure: Number (95% Confidence Interval); unit: Proportion of participants
Arm/Group | Arm A (Step 1: Internet-based Intervention; Step 2: Genetic Counseling Substudy) | Arm B (Step 1: Usual Care Control; Step 2: Genetic Counseling Substudy) | Arm C (Step 1: no Participation; Step 2: Genetic Counseling Substudy)
Number analyzed (Participants) | 7 | 4 | 7
Proportion of participants | 0.43 [0.10 to 0.82] | 0.5 [0.07 to 0.93] | 0.71 [0.29 to 0.96]

6. Primary Outcome: Proportion of Participants Who Complete Germline Testing in the Genetic Counseling Substudy (Step 2)
Description: as for outcome 5
Time Frame: Assessed at baseline at Step 2
Population: Eligible patients who agreed to participate in Step 2 genetic counseling substudy
Measure: Number (95% Confidence Interval); unit: Proportion of participants
Arm/Group | Arm A (Step 1: Internet-based Intervention; Step 2: Genetic Counseling Substudy) | Arm B (Step 1: Usual Care Control; Step 2: Genetic Counseling Substudy) | Arm C (Step 1: no Participation; Step 2: Genetic Counseling Substudy)
Number analyzed (Participants) | 7 | 4 | 7
Proportion of participants | 0.43 [0.10 to 0.82] | 0.25 [0.01 to 0.81] | 0.57 [0.18 to 0.90]

7. Secondary Outcome: Change of Scores on Cancer Genetic Knowledge Scale From Baseline to Post-genetic Education by Arm and Sex
Description: There are 14 items in the questionnaire of Cancer Genetic Knowledge Scale. The total score ranges between 14 and 70. Higher scores indicate more/better knowledge. The questionnaire was administered at baseline and post-genetic education. The change of scores from baseline to post-genetic education were calculated and interaction between arm and sex was evaluated.
Time Frame: Assessed at baseline and post-genetic education (about 1-2 weeks post-baseline)
Population: Eligible patients who completed both baseline and post-genetic education questionnaires were included in the analysis.
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Arm A (Step 1: Internet-based Intervention) | Arm B (Step 1: Usual Care Control)
Number analyzed (Participants) | 184 | 178
score on a scale
  Male: number analyzed (Participants) | 75 | 83
  Male | 1.4 (4.0) | -0.5 (3.7)
  Female: number analyzed (Participants) | 109 | 95
  Female | 1.5 (4.5) | -1.1 (3.6)

8. Secondary Outcome: Change of Scores on Patient-Reported Outcomes Measurement Information System (PROMIS) - Depression From Baseline to Post-genetic Education by Arm and Sex
Description: There are 4 items in the PROMIS - Depression questionnaire. The total score ranges between 4 and 20. Higher scores indicate more depression. The questionnaire was administered at baseline and post-genetic education. The change of scores from baseline to post-genetic education were calculated and interaction between arm and sex was evaluated.
Time Frame: Assessed at baseline and post-genetic education (about 1-2 weeks post-baseline)
Population: Eligible patients who completed both baseline and post-genetic education questionnaires were included in the analysis.
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Arm A (Step 1: Internet-based Intervention) | Arm B (Step 1: Usual Care Control)
Number analyzed (Participants) | 195 | 193
score on a scale
  Male: number analyzed (Participants) | 76 | 91
  Male | 0.2 (2.5) | 0 (2.3)
  Female: number analyzed (Participants) | 119 | 102
  Female | 0.2 (2.3) | -0.6 (2.6)

9. Secondary Outcome: Change of Scores on Patient-Reported Outcomes Measurement Information System (PROMIS) - Anxiety From Baseline to Post-genetic Education by Arm and Sex
Description: There are 4 items in the PROMIS - Anxiety questionnaire. The total score ranges between 4 and 20. Higher scores indicate more anxiety. The questionnaire was administered at baseline and post-genetic education. The change of scores from baseline to post-genetic education were calculated and interaction between arm and sex was evaluated.
Time Frame: Assessed at baseline and post-genetic education (about 1-2 weeks post-baseline)
Population: Eligible patients who completed both baseline and post-genetic education questionnaires were included in the analysis.
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Arm A (Step 1: Internet-based Intervention) | Arm B (Step 1: Usual Care Control)
Number analyzed (Participants) | 202 | 201
score on a scale
  Male: number analyzed (Participants) | 78 | 93
  Male | -0.3 (2.4) | -0.4 (1.9)
  Female: number analyzed (Participants) | 124 | 108
  Female | -0.3 (2.3) | -0.6 (2.5)

10. Secondary Outcome: Change of Scores on Impact of Events Scale (IES) From Baseline to Post-genetic Education by Arm and Sex
Description: There are 14 items in the questionnaire of Impact of Events Scale (IES). The total score ranges between 0 and 70. Higher scores indicate more stress. The questionnaire was administered at baseline and post-genetic education. The change of scores from baseline to post-genetic education were calculated and interaction between arm and sex was evaluated.
Time Frame: Assessed at baseline and post-genetic education (about 1-2 weeks post-baseline)
Population: Eligible patients who completed both baseline and post-genetic education questionnaires were included in the analysis.
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Arm A (Step 1: Internet-based Intervention) | Arm B (Step 1: Usual Care Control)
Number analyzed (Participants) | 183 | 191
score on a scale
  Male: number analyzed (Participants) | 76 | 87
  Male | -0.9 (8.6) | -1.5 (10.3)
  Female: number analyzed (Participants) | 107 | 104
  Female | -2.4 (10) | 0.9 (9.4)

11. Other Pre Specified Outcome: Factors Associated With Uptake of Remote Genetic Counseling in the Genetic Counseling Substudy (Step 2)
Description: The associations between patient characteristics and whether a patient receives genetic counseling will be evaluated.
Time Frame: Assessed at baseline in Step 2
Reporting Status: Not Posted

12. Other Pre Specified Outcome: Cognitive and Affective Responses to Confirmatory Germline Testing (Step 2)
Description: Cognitive and affective responses to confirmatory germline testing in advanced cancer patients with potential clinically significant incidental germline mutation identified in tumor profiling will be evaluated.
Time Frame: Assessed at baseline, within 3 days of remote genetic counseling, within 3 days of germline testing results received, and 3 months after germline testing results received in Step 2
Reporting Status: Not Posted

13. Other Pre Specified Outcome: Satisfaction and Regret/Disappointment Related to Tumor Genetic Test Results
Description: Satisfaction and regret/disappointment related to tumor genetic test results will be evaluated.
Time Frame: Assessed within 3 days of tumor test results received
Reporting Status: Not Posted

14. Other Pre Specified Outcome: How to Better Deliver Tumor Genetic Test Results and Germline Information in the Future
Description: How to better deliver tumor genetic test results and germline information in the future will be evaluated.
Time Frame: Assessed at baseline, within 3 days of genetic test results received, within 3 days of germline testing results received
Reporting Status: Not Posted

15. Other Pre Specified Outcome: Behavioral Responses to Confirmatory Germline Testing
Description: Behavioral responses (communication to others) to confirmatory germline testing in advanced cancer patients with potential clinically significant incidental germline mutation identified in tumor profiling will be evaluated.
Time Frame: as for outcome 12
Reporting Status: Not Posted

16. Other Pre Specified Outcome: Satisfaction and Regret/Disappointment Related to Genetic Counseling Service or Germline Genetic Test Results
Description: Satisfaction and regret/disappointment related to genetic counseling service or germline genetic test results will be evaluated
Time Frame: as for outcome 12
Reporting Status: Not Posted

ADVERSE EVENTS:
Time Frame: Adverse event data were not collected on this study.
Description: Adverse event data were not collected on this study.
Arm/Group | Arm A (Step 1: Internet-based Intervention; Step 2: Genetic Counseling Substudy) | Arm B (Step 1: Usual Care Control; Step 2: Genetic Counseling Substudy) | Arm C (Step 1: no Participation; Step 2: Genetic Counseling Substudy)
All-Cause Mortality (participants affected / at risk) | 0/0 | 0/0 | 0/0
Serious Adverse Events (participants affected / at risk) | 0/0 | 0/0 | 0/0
Other Adverse Events (participants affected / at risk) | 0/0 | 0/0 | 0/0

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: embargo of 60 days or less

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2019-05-14): https://cdn.clinicaltrials.gov/large-docs/52/NCT02823652/Prot_SAP_000.pdf